CLINICAL TRIAL: NCT01218451
Title: A Phase 3b, Randomized, Open Label, Feasibility Study of a Single Priming Dose of Meningococcal Group C Conjugate Vaccine (NeisVac-C) in Infants
Brief Title: NeisVac-C Single Prime Study in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 670901
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neisseria Meningitidis
MeSH Terms: interventions — 13-valent pneumococcal vaccine; Pentetic Acid; Hepatitis B Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Single dose of NeisVac-C vaccine at 4 months of age - Concomitant vaccinations of Infanrix hexa (0.5 mL) and Prevenar 13 (0.5 mL) at 2, 4 and 6 months of age - Booster vaccination with NeisVac-C, Infanrix hexa and Prevenar between 12 and 13 months of age
  Interventions: Biological: Meningococcal group C polysaccharide conjugate vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine
- Group 2 (Experimental): Single dose of NeisVac-C vaccine at 6 months of age - Concomitant vaccinations of Infanrix hexa (0.5 mL) and Prevenar 13 (0.5 mL) at 2, 4 and 6 months of age - Booster vaccination with NeisVac-C, Infanrix hexa and Prevenar between 12 and 13 months of age
  Interventions: Biological: Meningococcal group C polysaccharide conjugate vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine
- Group 3 (Active Comparator): Two doses of NeisVac-C vaccine at 2 and 4 months of age - Concomitant vaccinations of Infanrix hexa (0.5 mL) and Prevenar 13 (0.5 mL) at 2, 4 and 6 months of age - Booster vaccination with NeisVac-C, Infanrix hexa and Prevenar between 12 and 13 months of age
  Interventions: Biological: Meningococcal group C polysaccharide conjugate vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine

INTERVENTIONS:
Biological: Meningococcal group C polysaccharide conjugate vaccine — 0.5 mL dose, subcutaneous administration in right anterolateral thigh
  Other Names: NeisVac-C
Biological: Pneumococcal 13-valent conjugate vaccine — 0.5 mL dose, subcutaneous administration in right anterolateral thigh
  Other Names: Prevenar 13
Biological: Combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine — 0.5 mL dose, subcutaneous administration in right anterolateral thigh
  Other Names: Infanrix hexa

SUMMARY:
The purpose of this study is to assess the feasibility of a single priming dose of NeisVac-C in infants (at either 4 or 6 months of age), as determined by immune response.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an infant aged 8 to 11 weeks at the time of first vaccination
* Subject is clinically healthy as determined by the investigator's clinical judgment through collection of medical history and physical examination
* Subject was born at full term of pregnancy (>= 37 weeks) with a birth weight >= 2 kg
* The parent(s) or legally authorized representative of the subject provides written consent for participation
* The parent(s) or legally authorized representative of the subject has the ability to understand and comply with the requirements of the protocol
* The parent(s) or legally authorized representative and the subject will be available for the duration of the study
* The parent(s) or legally authorized representative of the subject agrees to keep a subject diary

Exclusion Criteria:

* Subject has a history of severe allergic reactions or anaphylaxis, or has a known sensitivity or allergy to any components of the vaccines
* Subject has had an acute or chronic infection requiring systemic therapy (antibiotic or antiviral) or other prescribed treatment within the 2 weeks prior to the first vaccination in this study
* Subject has a rash or dermatologic condition which may interfere with injection site reaction rating
* Subject currently has, or has a history of, any significant cardiovascular, respiratory, hepatic, renal, metabolic, autoimmune, rheumatic, hematological, neurological, or neurodevelopmental disorder
* Subject has a disease, or is currently undergoing a form of treatment, or was undergoing a form of treatment within 30 days prior to study entry, that could be expected to influence immune response
* Subject has received any blood products or immunoglobulins within 60 days of study entry
* Subject has received a live vaccine within 4 weeks or an inactivated or subunit vaccine within 2 weeks of the scheduled first vaccination
* Subject has previously been vaccinated against meningococcal C disease
* Subject has a known or suspected immune dysfunction
* Subject has a functional or surgical asplenia (e.g. due to a pathologic hemoglobinopathy, leukemia, lymphoma, etc.)
* Subject was administered an investigational drug within six weeks prior to study entry or is concurrently participating in a clinical study that includes the administration of an investigational product
* Subject or his/her parent(s) / legally authorized representative are in a dependent relationship with the study investigator or with a study team member; dependent relationships include close relatives (i.e. children, partner/spouse, siblings) as well as employees of the investigator or site conducting the study

Ages: 8 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 956 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with seroprotective antibody titers (rSBA titers >= 8) 1 month after completion of the primary vaccination in single-dose groups compared to the two-dose group | 1 month
Number of subjects with seroprotective antibody titers (rSBA titers >= 8) prior to the administration of the booster dose | 6 to 9 months (from 4-6 months of age until 12-13 months of age)
Number of subjects with seroprotective antibody titers (rSBA titers >= 128) 1 month after the administration of the booster dose | 1 month after booster dose (administered between 12-13 months of age)

SECONDARY OUTCOMES:
Antibody titers (rSBA) titers one month after completion of the primary vaccination | 1 month after primary vaccination
Antibody titers (rSBA titers) prior to the administration of the booster dose | Prior to booster dose
Antibody titers (rSBA titers)one month after the administration of the booster dose | 1 month after administration of booster dose
Frequency and severity of local and systemic ractions with onset within 3 days after each vaccination | Within 3 days after vaccination
Frequency and severity of adverse events observed during the entire follow up period | Entire follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Study Director — Baxter Healthcare Corporation
Locations (22):
- Poland (10):
  - NZOZ Vitamed, Bydgoszcz
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. Sw. Ludwika w Krakowie, Poradnia Pediatryczna Szczepien dla Dzieci z Grup Wysokiego Ryzyka, Krakow
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Oddzial Obserwacyjno-Zakazny dla Dzieci, Lodz
  - SP ZOZ Oddział Pediatyczny, Lubartów
  - Przychodnia Medycyny Wieku Rozwojowego, Poznan
  - NZLA Michałkowice Jarosz i partnerzy spolka lekarska, Siemianowice Śląskie
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - Szpital im. Świętej Jadwigi Śląskiej, Oddział Dziecięcy, Trzebnica
  - SPSK nr 1 we Wrocławiu, Klinika Pediatrii i Chorób Infekcyjnych, Wroclaw
  - NZOZ Zawidawie - Centrum Medyczne "Zatorska", Wroclaw
- Spain (12):
  - CSISP. Centro Superior de Investigación en Salud Pública, Almassora
  - CSISP. Centro Superior de Investigación en Salud Pública, Castellon
  - CSISP. Centro Superior de Investigación en Salud Pública, Catarroja
  - Hospital Universitario San Cecilio, Granada
  - CSISP. Centro Superior de Investigación en Salud Pública, L'Eliana
  - CSISP. Centro Superior de Investigación en Salud Pública, Puçol
  - CSISP. Centro Superior de Investigación en Salud Pública, Quart de Poblet
  - CSISP. Centro Superior de Investigación en Salud Pública, Sagunto
  - Instituto Hispalense de Pediatria, Seville
  - Hosptial Universitario Joan XXIII de Tarragona, Tarragona
  - CSISP. Centro Superior de Investigación en Salud Pública, Valencia
  - Hospital Comarcal Axarquía, Vélez-Málaga